CLINICAL TRIAL: NCT03602430
Title: Effect of Cholecalciferol on Hemodialysis Patients
Brief Title: Cholecalciferol on Hemodialysis Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona AlShahawey AlSayed Ghazy, Assistant lecturer of Clinical Pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: phCL 36
Record Dates: First submitted 2018-07-01; First posted 2018-07-26 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Hemodialysis Complication; Vitamin D Deficiency; Vascular Calcification
MeSH Terms: conditions — Vitamin D Deficiency; Vascular Calcification | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug Group (Experimental): twenty-five patients will receive 200.000 IU/month native vitamin D; (Cholecalciferol) orally in addition to their standard treatment for 3 months period
  Interventions: Drug: Cholecalciferol
- Placebo Group (Placebo Comparator): twenty-five patients will receive a placebo ampule with their standard treatment for 3 months period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Native vitamin D dose of 200IU to be given once per month to hemodialysis patients
  Other Names: Native vitamin D
  Arms: Drug Group
Drug: Placebo — A Placebo ampule will be given to hemodialysis patients once per month with their standard treatment for 3 months period. Same color, odor and size, only without the active constituent.
  Arms: Placebo Group

SUMMARY:
* Screening the prevalence of vitamin D deficiency among Egyptian hemodialysis patients on a single center (Ain Shams University hospital).
* Assessing the effect of the native type of vitamin D (Cholecalciferol) on replenishing its deficiency via extra-renal vitamin D receptors (VDR), among Egyptian hemodialysis patients.
* Assessing the effect of cholecalciferol on vascular calcification among Egyptian hemodialysis patients.
* Assessing the effect of cholecalciferol on Blood pressure, parathyroid hormone.

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes aged between 18-75 years
2. Patients on HD greater than 3 months at least.
3. Stable clinical condition (no hospitalization in the previous 3 months)
4. Informed consent in accordance with the Declaration of Helsinki.
5. PTH level between 150 - 800 pg/ml.

Exclusion Criteria:

1. Hypersensitivity to cholecalciferol.
2. Participant in an another clinical trial within the past 4 weeks.
3. Judged to be unsuitable as a subject by the attending physician.
4. Pregnant or breastfeeding female

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Vitamin D level | 3 months
  Target serum Vitamin D level ≥ 30 ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alshahawey M, El Borolossy R, El Wakeel L, Elsaid T, Sabri NA. The impact of cholecalciferol on markers of vascular calcification in hemodialysis patients: A randomized placebo controlled study. Nutr Metab Cardiovasc Dis. 2021 Feb 8;31(2):626-633. doi: 10.1016/j.numecd.2020.09.014. Epub 2020 Sep 21. PMID 33594986